CLINICAL TRIAL: NCT02332369
Title: EyeKon Medical, Inc. Capsular Tension Ring Clinical Study
Brief Title: EyeKon Medical Inc. Capsular Tension Ring Study
Acronym: CTR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: EyeKon Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EyeKon CTR--01
Record Dates: First submitted 2015-01-05; First posted 2015-01-06 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Cataract Extraction
Keywords: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Device (Experimental): Polymethylmethacrylate Capsular Tension Ring introduced into the posterior chamber of the eye following cataract surgery before the implantation of an intraocular lens.
  Interventions: Device: Capsular Tension Ring

INTERVENTIONS:
Device: Capsular Tension Ring

SUMMARY:
This study evaluates the safety and effectiveness of a capsular tension ring (CTR) when used during cataract surgery. Capsular Tension Rings are used during intraocular lens implantation to give added support in order to keep the intraocular lens well centered, especially in eyes with weak or partially absent zonules. In many cases, capsular tension rings allow a lens to be successfully implanted into an eye which otherwise could not have supported an intraocular lens.

DETAILED DESCRIPTION:
The clinical study of the CTR-10 and CTR-12 Capsular Tension Rings is to be conducted with the following objectives:

1. Determine the ability of the device to maintain the shape of the capsular bag and therefore keep the intraocular lens centered;
2. Determine post-operative visual acuity of patients receiving the capsular tension ring as a secondary method of determining the efficacy;
3. Describe the occurrence and time course of postoperative complications and adverse reactions for capsular tension ring implant subjects;
4. Describe the occurrence of postoperative complications for the implant group and their relationship to ocular complications.
5. Identify groups within the implant study population that are at "high risk" of particular complications.
6. Collect and analyze against those historical controls published by FDA data on:

   1. Overall Visual Acuity
   2. Best Case Visual Acuity
   3. Cumulative Hyphema
   4. Cumulative Macular Edema
   5. Cumulative Retinal Detachment
   6. Cumulative Pupillary Block
   7. Cumulative Lens Dislocation
   8. Cumulative Endophthalmitis
   9. Cumulative Hypopyon
   10. Cumulative Surgical Reintervention
   11. Persistent Macular Edema
   12. Persistent Corneal Edema
   13. Persistent Iritis
   14. Persistent Raised IOP Requiring treatment
   15. Frequency and degree of posterior capsule opacification

The investigational plan for the clinical study of capsular tension rings is designed to satisfy the requirements of the Investigational Device Exemption (IDE) regulations, which require a well-controlled clinical trial with ongoing monitoring to evaluate the safety and efficacy of the intraocular lenses.

The study will consist of adult patients who will be enrolled into the study. The results of these implants will be carefully monitored for approximately twelve (12) months.

ELIGIBILITY:
Inclusion Criteria:

* The patient is in good general and ocular health, having a vision-reducing cataract in the intended operative eye.
* The intended operative eye has a Snellen best corrected visual of 20/40 or worse for distance or the refraction worsens to this level with glare testing.
* The patients' worse seeing Eye is 20/70 or better.
* The patient is willing and able to complete all required postoperative visits.
* The patient is willing to sign a statement of informed consent.
* The patient is at least 21 years old.
* The patient requires cataract surgery with IOL implantation.
* The patient has observed or suspected weakened, torn, missing or otherwise compromised zonules (torn or missing estimated not to exceed one-third of the capsular bag diameter) due to Pseudoexfoliation Syndrome, Marfans Syndrome, trauma or other zonular compromising condition.
* The capsule is intact during insertion.

Exclusion Criteria:

* Only one functional eye
* Capsular bag tearing beyond the point where the surgeon thinks it is in the best interest of the patient to have a capsular ring implanted
* Significant zonular didlysis during surgery
* Preoperative ocular infection
* Ocular inflammation or uveitis
* Amblyopia
* Aniridia
* Congenital cataracts
* Cataracts due to rubella
* Corneal disease
* Diabetes
* Preoperative intraocular pressure over 21 mm Hg
* Iritis
* Iris atrophy
* Pseudophakic lens exchange
* Microphthalmia
* Optic atrophy
* Macular degeneration
* Retinal detachment
* Retinal degeneration
* Vitritis
* Flat anterior chamber
* Other conditions as noted by the surgeon which may compromise the safety of the patient or the accuracy of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2005-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | At all pre/post op CFR's for 1 year.
  Best case visual acuity at 1 year of follow-up based upon LogMar score.

SECONDARY OUTCOMES:
Adverse Events | 1 Year
  Adverse events will be compared to the FDA historical grid and must be less than or equal to those shown in the grid on a percentage of patients enrolled basis.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Robinson, Study Director — Sponsor/CEO
Locations (3):
- United States (3):
  - Stephenson Eye Associates, Venice, Florida
  - Comprehensive Eye Care Ltd., Washington, Missouri
  - Brazosport Eye Institute, Lake Jackson, Texas